CLINICAL TRIAL: NCT04637477
Title: Rush Coronavirus Disease Virtual Lifestyle Program to Boost Host Resistance in Patients With Elevated Cardiometabolic Risk: A Proof-of-Concept Study
Brief Title: Virtual Enhanced Lifestyle for Metabolic Syndrome (ELM) Proof-of-Concept Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: University of Missouri, Kansas City (Other); University of Colorado, Denver (Other); Geisinger Clinic (Other); Rochester Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20061108
Record Dates: First submitted 2020-11-06; First posted 2020-11-19 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Metabolic Syndrome; Obesity
Keywords: Lifestyle
MeSH Terms: conditions — Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual ELM (Experimental)
  Interventions: Behavioral: Virtual ELM

INTERVENTIONS:
Behavioral: Virtual ELM — Participants will attend 1.5-hour virtual group-based sessions for 12 weeks. The program includes physical activity, cooking demonstrations, and group discussions. All sessions are led by a registered dietitian and health psychologist.

SUMMARY:
This is a proof-of-concept study of a virtual version of a lifestyle intervention aimed at reducing cardiometabolic risk in patients with the Metabolic Syndrome (MetS). The aim is to recruit 12 patients at high risk for coronavirus infection based upon a diagnosis of obesity and the MetS, conduct a 12-week virtual version of the in-person intervention, and explore efficacy using clinically significant pre-specified targets for weight, diet, physical activity, stress, and markers of inflammation. In addition, the investigators will explore safety, fidelity, feasibility, and acceptability.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with components of the metabolic syndrome, defined by an adapted version of the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO (Alberti, 2009). Surrogates for waist circumference and fasting glucose were selected to help identify prospective participants using medical records. Participants must have ≥ 2 of the following five criteria to participate in the study:

   * Waist circumference based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women or BMI≥30
   * Triglycerides ≥150 mg/dL or treatment for elevated triglycerides
   * HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL
   * Systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or treatment for hypertension
   * Fasting plasma glucose 100-125 mg/dL (range inclusive), or on metformin, or HbA1c between 5.7 and 6.4.
2. Age 18 years or older
3. Highly motivated to make lifestyle changes as a way to manage the MetS.

Exclusion Criteria:

1. Individuals who report being unable to walk 2 consecutive blocks without assistance are ineligible. Additionally, individuals who endorse pain, tightness, or pressure in their chest during physical activity (on question 1 of the EASY screener) or current dizziness or lightheadedness (on question 2 of the EASY screener) may not be randomized without providing documentation in writing from their physician indicating that they have been cleared for participation in the trial.
2. Unwilling, unable, or not ready to make the lifestyle changes prescribed in ELM
3. BMI <27 or > 40
4. Weight > 397 lbs. The Fitbit Aria scale, utilized in the intervention, measures up to 397 lbs.
5. Unable to consistently attend group classes at the anticipated time due to schedule conflicts or other reasons.
6. Unable or unwilling to give an informed consent or communicate with study staff.
7. Unable or unwilling to complete accelerometer data collection.
8. Does not have reliable access to the internet.
9. Does not have a smart phone. Must be willing to download the Fitbit app on their smart phone.
10. Not fluent in English
11. Current diagnosis of type 1 or type 2 diabetes, on any diabetes medications except metformin, or has a screening A1c ≥6.5
12. Inpatient treatment for a psychiatric condition within the past 6 months, or currently receiving treatment for schizophrenia or other serious psychiatric illness
13. Probable major depression, defined as a PHQ-8 score ≥10
14. Pregnant women, planning a pregnancy in the next 2 months, given birth in the last 6 months, or currently breastfeeding
15. ≥ 30 total days of oral corticosteroid use within the last year, history of solid organ transplant, or history of stem cell transplant
16. Problematic use of alcohol and/or recreational drugs, defined as ASSIST screening score of ≥27.
17. Self-reported or known history of an eating disorder (e.g., binging and purging) in the past 5 years
18. Use of weight loss medications (Qsymia, orlistat, phentermine, Saxenda, etc.) in the last 3 months, or unwilling to abstain from taking weight loss medications or supplements during the trial
19. History of bowel resection surgery or bariatric surgery
20. Any medical condition known to influence the etiology of MetS as judged by the study physician (e.g., uncontrolled hypothyroidism, endocrine hypertension, etc)
21. History of major cardiovascular illness, including: a) stroke; b) myocardial infarction; c) congestive heart failure requiring hospitalization, or greater than NYHA heart failure class I; d) uncontrolled hypertension (SBP>180 or DBP > 109); e) unstable angina or an active prescription for sublingual nitroglycerin; or f) other major cardiovascular illness which the site PI determines could limit ability to participate in the trial. Individuals screened for participation, whose screening systolic blood pressure is ≥160 and ≤179, or whose screening diastolic blood pressure is ≥100 and ≤109 are considered to have MODERATE, or Stage 3 Hypertension. If they otherwise qualify and wish to participate in ELM, they will be referred to their physician for clearance prior to randomization.
22. Cognitive impairment
23. Visual or hearing impairment
24. Currently taking or expecting to take any of the following exclusionary medications:

    1. Antiretroviral therapy (e.g., HAART)
    2. Weight loss medications (as in #14)
    3. Medications known to significantly influence weight or metabolic outcomes
    4. Diabetes drugs other than metformin (as in #7)
25. Receiving dialysis
26. Cancer treatment within the last 6 months, excluding chemoprophylaxis or treatment for non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Fifty percent of participants will lose >5% of baseline weight after completing the intervention at 3 months. | 3 months after baseline assessment
  Weight is recorded in kilograms to the nearest 0.1 kg using a flat scale.

SECONDARY OUTCOMES:
Remission of components of metabolic syndrome | Measured at 3 months from baseline
  The proportion of participants who are in remission of the metabolic syndrome (MetS) at 3 months will be calculated. MetS is defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO as having 3 or more risk factors for cardiovascular disease. To be considered in remission of MetS the participant must have less than 3 of the following 5 criteria: 1) Waist circumference based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women; 2) Fasting triglycerides ≥150 mg/dL or treatment for elevated triglycerides; 3) Fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL; 4) Systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or treatment for hypertension; and 5) Fasting plasma glucose 100-125 mg/dL.
Vegetable consumption | Measured at 3 months from baseline
  The proportion of participants who eat 2 cups of vegetables per day. This will be assessed using the National Cancer Institute (NCI) Fruit and Vegetable Intake Screener from the Eating at America's Table Study: All Day Screener.
Physical activity | Measured at 3 months from baseline
  The proportion of participants who achieve 150 minutes of at least moderate intensity physical activity per week will be calculated. Activity is measured using an accelerometer (Actigraph wGT3X-BT) worn on the right hip for 7 days and for at least 10 hours/day.
Facets of Mindfulness | Measuring change from baseline mindfulness at 3 months
  Participants will complete the Five Facet Mindfulness Questionnaire. A subscale comprised of 3-facets (observe, act with awareness, and nonreact) will be utilized to measure mindfulness in ELM. The proportion of participants who improve in a 3-facet mindfulness score of greater than or equal to 1 standard deviation of baseline distribution will be calculated. The scale range for the 5-facet mindfulness questionnaire is 39-195 with a lower score reflecting less mindfulness. The 3-facet scale range is 23-115 with a lower score reflecting less mindfulness.
Habit formation | Measured at 3 months after baseline
  The proportion of participants who improve in habit strength in 4 domains (diet, physical activity, emotional control, and sensory awareness), defined as a mean of ≥ 4 on the Self-Report Habit Index will be calculated. A 5-point Likert scale will be used with a scale range from 0 to 20. A lower score reflects a weaker habit.

OTHER OUTCOMES:
Metabolic syndrome severity score | Measured at 3 months after baseline
  MetS components will be assessed as a continuous sex- and race/ethnicity-specific score. The higher the MetS Severity score, the higher risk/severity. (Gurka MJ, Lilly CL, Oliver MN, DeBoer MD. An examination of sex and racial/ethnic differences in the metabolic syndrome among adults: a confirmatory factor analysis and a resulting continuous severity score. Metabolism. 2014;63:218-25).
Weight loss | Measuring change from baseline to 3 months
  Calculate the average weight loss (kg). Weight is recorded in kilograms to the nearest 0.1 kg using a flat scale.
Blood pressure (metabolic syndrome component) | Measured at baseline and 3 months
  The percent of participants with the blood pressure component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria for blood pressure is met when systolic blood pressure ≥130 m Hg, diastolic blood pressure ≥85 mm Hg, or self-reported treatment for hypertension.
  Average of 3 seated resting blood pressure measurements using NHANES protocol and cuff sizes based on arm circumference. Device is OMRON HEM-907XL
  Cuff sizes:
  Small (17.0-22.0 cm) Medium/Adult (22.1-32.0 cm) Large (32.1-42.0 cm) Extra Large (42.0-50.0 cm)
Waist circumference (metabolic syndrome component) | Measured at baseline and 3 months
  Percent of participants with the waist circumference component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria is based on AHA/NHLBI (ATP III) cut points of ≥ 102 cm for men and ≥ 88 cm for women.
  Waist circumference will be measured using a tape measure, following the National Heart, Lung, and Blood Institute waist circumference assessment guidelines.
Triglycerides (metabolic syndrome component) | Measured at baseline and 3 months
  The percent of participants with the triglyceride component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria for elevated triglyceride levels are fasting triglycerides ≥150 mg/dL or treatment for elevated triglycerides.
  A fasting blood sample will be sent to Quest diagnostics for analysis.
High-Density Lipoproteins (HDL) cholesterol (metabolic syndrome component) | Measured at baseline and 3 months
  The percent of participants with the HDL cholesterol component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. The criteria for low HDL are fasting HDL cholesterol <40 mg/dL in men or <50 mg/dL in women, or treatment for low HDL.
  A fasting blood sample will be sent to Quest diagnostics for analysis.
Fasting plasma glucose (metabolic syndrome component) | Measured at baseline and 3 months
  The percent of participants with the fasting glucose component of the Metabolic Syndrome as defined by the Joint Interim Statement of the IDF, NHLBI, AHA, WHF, IAS, IASO. Fasting plasma glucose 100-125 mg/dL (range inclusive) is considered a component of the metabolic syndrome. A fasting blood sample will be sent to Quest diagnostics for analysis.
Body mass index | Measuring change from baseline to 3 months
  The percent of participants who lowered their Body Mass Index (BMI). Height will be recorded in cm to nearest 0.25 cm and weight recorded in kg to nearest 0.1 kg. BMI = weight (kg) / height squared (m). The weight and height will be combined to report BMI in kg/m^2.
Frequency of contacts within health network | Measuring change from baseline to 3 months
  The frequency of contacts within participants' health network.
Energy and vitality index | Measuring change from baseline to 3 months
  Percent of participants who improved in the energy and vitality subscale from the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) version 1. The scale range is 0 to 100 with a low score reflecting a lower energy and vitality.
Perceived stress | Measuring change from baseline to 3 months
  Measuring change of perceived stress score from baseline using the 10-item Perceived Stress Scale. The scale range is from 0 to 40. A lower score reflects lower levels of stress.
Depressive symptoms | Measuring change from baseline to 3 months
  Measuring change of depressive symptoms from baseline using the 8-item self-report Patient Health Questionnaire Depression Scale (PHQ-8). This scale ranges from 0 to 24 with a lower score reflecting less (or no) depressive symptoms.
Hemoglobin A1c levels | Measuring change from baseline to 3 months
  Measuring change in Hemoglobin A1c levels. A blood assay will be analyzed by Quest Diagnostics. Standard safety procedures are used in performing the participant blood draw required for this measure.
Sugar-sweetened beverages | Measuring change from baseline to 3 months
  Measuring change in frequency of consumption of sugar-sweetened beverages using the Behavioral Risk Factor Surveillance System - Beverage Items.
Eating competence | Measuring change from baseline to 3 months
  Measuring change on eating competence using the 16-item Eating Competence Survey. The scale ranges from 0 to 48 with a higher score reflecting a better outcome.
C-reactive protein (hs-CRP) | Measuring change from baseline to 3 months
  Measuring decrease inflammation by using the benchmark of 20% improvement in hs-CRP.
Interleukin 6 (IL-6) | Measuring change from baseline to 3 months
  Measuring decrease inflammation by using the benchmark of 20% improvement in IL-6.
Fidelity of intervention | Measuring during 3-month lifestyle program
  Explore the fidelity of treatment delivery, receipt, and enactment. Treatment delivery is measured by the investigator reviewing the session recordings and completing a standardized form assessing the interventionists' ability to deliver the program as designed. Receipt of treatment is assessed by attendance. Enactment of treatment is self-reported by participants in a 4-item questionnaire after each session.
Feasibility of recruitment | Up to 12 weeks
  Explore feasibility of recruitment by reviewing the screened to enrollment ratio. Research staff will also take qualitative notes on the process to inform future recruitment strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Powell, PhD, Principal Investigator — Rush University Medical Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - University of Missouri-Kansas City School of Medicine, Kansas City, Missouri